CLINICAL TRIAL: NCT00363792
Title: The Effect of Glyceryl Trinitrate and Diamox on Blood-Oxygenation-Level-Dependent.Signal (BOLD-Signal) and Cerebral Haemodynamics With the Use of a 3-Tesla MRI-Scan.
Brief Title: Effect of GTN and Diamox Measured by BOLD-Response.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Headache Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: KA-20060085
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2006-08

CONDITIONS: Healthy
Keywords: Healthy subjects
MeSH Terms: interventions — Nitroglycerin

INTERVENTIONS:
Drug: Glyceryl trinitrate, azetazolamide

SUMMARY:
In healthy subjects different cerebral haemodynamic values wished to be determined after infusion of the NO donor Glyceryl trinitrate (GTN) and Diamox. The different values we wish to determine are:

* Blood-oxygenation-level-Dependent-signal (BOLD-signal) after visual stimulation.
* Changes in the diameter of a. cerebri media.
* Changes in the regional and global cerebral blodd flow (CBF) with the help of the arterial Spin labeling (ASL) method.

DETAILED DESCRIPTION:
Experimental headache models give a unike opportunity to study pathophysiological mechanisms of prim. headache types such as migraine. Previous studies have used different methods that have had limitations and none of them have had the opportunity to study neuronal activation. But that is possible with the application of functional magnetic resonance (fMRI).

Before we apply fMRI to our experimental headache models it is needed to determine how the BOLD response is influenced and changed by the infusion of different drugs such as the NO donor Glyceryl Trinitrate (GTN) and Diamox (acetazolamide). It is known that GTN causes dilation of the cerebral arteries without having any effect on the regional cerebral blood flow. It is not known what effect GTN has on the BOLD response. Diamox (azetazolamide) increases the CBF but it is uncertain what effect the drug has on the BOLD response. Previous studies disagree gravely on this point.

In this study we will be giving infusion of GTN and Diamox in healty subjects to determine:

* Blood-oxygenation-level-Dependent-signal (BOLD-signal) after visual stimulation.
* Changes in the diameter of a. cerebri media.
* Changes in the regional and global cerebral blodd flow (CBF) with the help of the arterial Spin labeling (ASL) methode.

For the study we will be using a 3-Tesla MRI-scan.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* age 18-55 years
* weight 50-100 kg

Exclusion Criteria:

* Tension type headache more the once per month.
* other types of headache
* Daily use of medication other the birthcontrol pills.
* Pregnant or lactating women.
* headache on the examination date.
* contraindications to MRI-scan.
* hypotension or hypertension.
* mental illness og substance abuse.
* other significant conditions determined by the examining doctor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Study Completion 2007-05

PRIMARY OUTCOMES:
Changes in BOLD response
Changes in a. cerebri media diameter
Changes in CBF

SECONDARY OUTCOMES:
headache score

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, MD, Phd,, Study Chair — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark